CLINICAL TRIAL: NCT04439708
Title: Biomarkers Analysis of Mineralocortoid Receptor Activation in the Serum and Ocular Fluid of Patients With Choroidal Neovascularization
Brief Title: Biomarkers and Choroidal Neovascularization
Acronym: BioNéoRet
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C18-08; 2018-A02099-46 (Registry Identifier: 2018-A02099-46)
Record Dates: First submitted 2020-03-02; First posted 2020-06-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Choroidal Neovascularization; Mineralocorticoid Excess
Keywords: central serous chorioretinopathy; age related macular degeneration; biomarker
MeSH Terms: conditions — Choroidal Neovascularization; Hyperaldosteronism; Central Serous Chorioretinopathy; Macular Degeneration | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and aqueous humor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients with choroidal neovascularization in the context of age-related macular degeneration or central serous chorioretinopathy
  Interventions: Other: Blood and aqueous humor biomarker of treatment response
- Group 2: Control group : patients without choroidal neovascularization
  Interventions: Other: Blood and aqueous humor biomarker of treatment response

INTERVENTIONS:
Other: Blood and aqueous humor biomarker of treatment response — Blood analyses and aqueous humor analysis

SUMMARY:
The aim of the study is to find biomarkers in the blood and aqueous humor of patients with type 1 choroidal neovascularization and correlate them with the response to anti-VEGF treatment.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the most frequent cause of blindness in industrialized countries. Multiple molecular pathways have been implicated in the pathogenesis of choroidal neovascularization (CNV). Currently, the treatment relies on neutralization of VEGF (Vascular Endothelial Growth Factor). However some patients have an incomplete response to anti-VEGF treatment. A recent study suggested the implication of the mineralocorticoid receptor pathway in the formation of CNV.

The study (of investigators) aim is to evaluate the concentation of metabolites of MR pathway in the blood and aqueous humor of patients with CNV and compared them with patients without CNV in order to increase our understanding of CNV pathogenesis and find potential biomarker of response to anti-VEGF treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients of group 1:

* Patients with type 1 choroidal neovascularization in a context of central serous chorioretinoathy or age related macular degeneration
* Patients without intravitreal injection or last intravitreal injection > 3 months
* Informed signed consent

Patients of group 2:

* Patients without choroidal neovascularization
* Patients with intraocular surgery (cataract or vitrectomy surgery)
* Signed consent

Exclusion Criteria:

* Myocardial infarction < 12 months
* Chronic renal failure
* Inflammatory disease
* Infectious disease :HIV, viral hepatitis, tuberculosis
* Type 1 or 2 Diabetes
* Patients treated by mineralocorticoid antagonist treatment.
* Type 2 or 3 choroidal neovascularization
* Pregnant woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1 : patients with type 1 choroidal neovascularization Group 2: patients without choroidal neovascularization before ocular surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
biomarker analysis in blood and aqueous humor of patients with neovascularization and controls | 24 months
  Biomarker concentrations (pg/ml) will be evaluated with ELISA (Enzyme Linked ImmunoSorbent Assay).
biomarker analysis in blood and aqueous humor of patients with neovascularization and controls | 24 months
  Biomarker concentrations (pg/ml) will be evaluated with Mulitplex Biorad.

SECONDARY OUTCOMES:
biomarkers and treatment response | 24 months
  Correlation between biomarker level and the response to anti-VEGF treatment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ophtalmopole Hôpital Cochin, Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Background] Suzuki M, Nagai N, Izumi-Nagai K, Shinoda H, Koto T, Uchida A, Mochimaru H, Yuki K, Sasaki M, Tsubota K, Ozawa Y. Predictive factors for non-response to intravitreal ranibizumab treatment in age-related macular degeneration. Br J Ophthalmol. 2014 Sep;98(9):1186-91. doi: 10.1136/bjophthalmol-2013-304670. Epub 2014 Apr 7. PMID 24711658
- [Background] Kersten E, Paun CC, Schellevis RL, Hoyng CB, Delcourt C, Lengyel I, Peto T, Ueffing M, Klaver CCW, Dammeier S, den Hollander AI, de Jong EK. Systemic and ocular fluid compounds as potential biomarkers in age-related macular degeneration. Surv Ophthalmol. 2018 Jan-Feb;63(1):9-39. doi: 10.1016/j.survophthal.2017.05.003. Epub 2017 May 15. PMID 28522341
- [Background] Rezar-Dreindl S, Sacu S, Eibenberger K, Pollreisz A, Buhl W, Georgopoulos M, Krall C, Weigert G, Schmidt-Erfurth U. The Intraocular Cytokine Profile and Therapeutic Response in Persistent Neovascular Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2016 Aug 1;57(10):4144-50. doi: 10.1167/iovs.16-19772. PMID 27537264
- [Background] Zhao M, Mantel I, Gelize E, Li X, Xie X, Arboleda A, Seminel M, Levy-Boukris R, Dernigoghossian M, Prunotto A, Andrieu-Soler C, Rivolta C, Canonica J, Naud MC, Lechner S, Farman N, Bravo-Osuna I, Herrero-Vanrell R, Jaisser F, Behar-Cohen F. Mineralocorticoid receptor antagonism limits experimental choroidal neovascularization and structural changes associated with neovascular age-related macular degeneration. Nat Commun. 2019 Jan 21;10(1):369. doi: 10.1038/s41467-018-08125-6. PMID 30664640